CLINICAL TRIAL: NCT01885767
Title: Neurofibromatosis (NF) Registry Portal Funded by Children's Tumor Foundation
Brief Title: Neurofibromatosis (NF) Registry Portal
Status: Recruiting | Type: Observational
Sponsor: The Children's Tumor Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CTF001
Record Dates: First submitted 2013-05-22; First posted 2013-06-25 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Neurofibromatosis 1; Neurofibromatosis 2; Schwannomatosis
Keywords: Neurofibromatosis; NF; Neurofibromatosis 1; NF1; Neurofibromatosis 2; NF2; Schwannomatosis
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatosis 2; Schwannomatosis; Neurofibromatoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- NF1: Patients meeting clinical and/or genetic criteria for Neurofibromatosis 1
- NF2: Patients meeting clinical and/or genetic criteria for Neurofibromatosis 2
- SchW: Patients meeting clinical and/or genetic criteria for Schwannomatosis

SUMMARY:
The NF Registry is a database of patient-reported symptoms, treatments, and experiences with their neurofibromatosis disease. It is a contact registry to relay clinical trial opportunities to targeted patient subgroups, and to supply de-identified disease data to researchers. It has the potential to become a natural history resource.

DETAILED DESCRIPTION:
Patients and parents of patients will be made aware of the Neurofibromatosis (NF) Registry through various non-commercial information sources such as the Children's Tumor Foundation (CTF) website, CTF-affiliated NF clinics, social media, CTF educational and fundraising events, and other nonprofit organizations and foundations such as the National Organization for Rare Diseases (NORD) and social media.

The NF Registry will be accessed by individual adult (over age 18) subjects via a web-based patient portal. The portal contains an IRB-approved informed consent form. Following consent, the registrant creates an account which is activated after email confirmation. An account can be created by an adult patient with the disorder, or by the parent or guardian of a child with the disorder. Account creators are required to enter identifiable contact and demographic data.

After the account is created, the account owner enrolls themselves or a minor family member (or both) and completes an on-line survey. There are separate surveys for NF1, NF2, and Schwannomatosis. The surveys ask about about the affected individual's medical and family history of the disease, testing and diagnosis, clinical manifestations (e.g., tumor types and locations) interventions and therapies, and quality of life. The account holder chooses whether to receive emails from the Registry with information about relevant clinical trials and studies for which they may be eligible.

Participant's responses are used to compile charts and graphics of de-identified aggregate data. Registered patients may view this data. Researchers may apply to our Data Use Committee for access to de-identified data or for subject recruitment emails to be sent to specific patient subgroups. Data capture and security for the NF Registry is done under contract by OpenApp (Dublin, Ireland), a web-based patient opt-in registry provider.Participants will be asked to update their information at least once a year. Their information will be stored in the NF Registry for an indefinite period of time. This longitudinal study is intended as a resource for patients and researchers. There is no specific outcome measure or anticipated endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with NF1
* Diagnosed with NF2
* Diagnosed with Schwannomatosis

Exclusion Criteria:

* Failure to complete account registration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected with NF1, NF2, or Schwannomatosis
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2012-06; Primary Completion 2030-06 (Estimated); Study Completion 2050-06 (Estimated)

PRIMARY OUTCOMES:
To create a natural history of NF1, NF2, and schwannomatosis | final report in 2050 with descriptive statistics
  patients will input medical information and treatment information about their NF and update at least yearly in an ongoing natural history study

CONTACTS AND LOCATIONS:
Overall Officials: Kate Kelts, B.S.N., Principal Investigator — The Children's Tumor Foundation
Locations (1):
- Children's Tumor Fundation, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
deidentified data only may be shared

REFERENCES:
- See also: NF Registry — https://nfregistry.org